CLINICAL TRIAL: NCT02238821
Title: Role of the MET Oncogene in Human Colorectal Cancer. Possible Implications in the Activation of an Acquired Pro-thrombotic Condition - A Translational Study
Brief Title: Role of the MET Oncogene in Human Colorectal Cancer - A Translational Study
Acronym: COMET
Status: Completed | Type: Observational
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: MET/colon 06
Record Dates: First submitted 2014-09-01; First posted 2014-09-12 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: resectable colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- resectable colorectal cancer

SUMMARY:
The MET oncogene is known to sustain the Trousseau's syndrome in murine experimental models, featuring association of carcinogenesis with a blood procoagulant disorder. MET is frequently overexpressed in colorectal cancer, a tumor where venous thromboembolism (VTE) may occur in association with poor prognosis, but the biological and genetic factors that cause VTE are still obscure.

The Investigators propose to study whether in patients harboring a surgically resectable colorectal cancer the MET oncogene is expressed and may be associated with a blood thrombophilic condition that favors the onset of VTE.

These data would have two main implications: (i) for the first time, a direct genetic link between the MET oncogene and a procoagulant disorder would be demonstrated in humans; (ii) the procoagulant alterations would have diagnostic/prognostic significance for the identification of patients at risk for poor outcome, and implementation of appropriate therapeutic protocols.

ELIGIBILITY:
Inclusion Criteria:

* age > or = 18;
* age < or = 80;
* Clinical diagnosis of colorectal tumor by CT, MRI or endoscopy;
* surgically resectable tumor;

Exclusion Criteria:

* Inclusion in other clinical protocols requiring administration of anticoagulant drugs;
* Life expectancy < 6 month;
* Clinical diagnosis of thrombophilic condition by laboratory analysis;
* Previously implanted Central Venous Catheter;
* Previous or concomitant second neoplasia;
* Clinical diagnosis of kidney, liver or heart failure;
* Inflammatory markers alteration associated with disease unrelated to neoplasia (infection, connective tissue disease etc);
* Severe hemostasis disorder;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resectable colorectal tumor with survival prognosis>6 month
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-10; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Scoring MET expression in colorectal tissue sections by immunohistochemical analysis | After surgical resection of the tumor, approximately 3-5 days after enrollement
Scoring the expression of Plasminogen Activator Inhibitor -1 in colorectal cancer tissue sections by Immunohistochemical analysis | After surgical resection of the tumor, approximately 3-5 days after enrollement
Scoring the expression of COX-2 in colorectal cancer tissue sections by Immunohistochemical analysis | After surgical resection of the tumor, approximately 3-5 days after enrollement

CONTACTS AND LOCATIONS:
Overall Officials: Paolo M Comoglio, MD, Study Director — Fondazione del Piemonte per l'Oncologia
Locations (1):
- Fondazione del Piemonte per l'Oncologia, Candiolo, TO, Italy